CLINICAL TRIAL: NCT05285696
Title: A Phase 1 Study to Evaluate the Safety and Dosimetry of [68Ga]-NOTA-hGZP (CSB-111) PET Imaging in Healthy Human Volunteers.
Brief Title: Study to Evaluate the Safety and Dosimetry of [68Ga]-NOTA-hGZP (CSB-111) PET Imaging in Healthy Human Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytosite Biopharma Inc. (Industry)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CYT-002-01
Record Dates: First submitted 2021-10-28; First posted 2022-03-17 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [68Ga]-NOTA-hGZP (CSB-111) Injection (Experimental): Eligible participants will receive a single IV injection of CSB-111 up to 40 micro grams
  Interventions: Drug: CSB-111

INTERVENTIONS:
Drug: CSB-111 — [68Ga]-NOTA-hGZP is a PET imaging agent.
  Other Names: [68Ga]-NOTA-hGZP

SUMMARY:
Phase one study to evaluate the safety and dosimetry of [68Ga]-NOTA-hGZP (CSB-111) PET Imaging in healthy human volunteers.

DETAILED DESCRIPTION:
This study aims to assess the safety and evaluate the dosimetry of CSB-111. This study will estimate organ dosimetry and the overall effective dose, a requirement for expanding the human use of a radiopharmaceutical.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy participants aged between 18 and 65 years old.
2. For females of childbearing potential, a negative serum or urine beta-human chorionic gonadotropin (β-hCG) pregnancy test must be obtained at the day of the procedure prior to CSB-111 administration.
3. Willing and able to undergo all study procedures.
4. Willing and able to understand the written informed consent and sign the consent document prior to any study-related procedure.
5. Willing to refrain from strenuous exercise for the 24 hours prior to CSB-111 administration

Exclusion Criteria:

1. History of allergic reactions to compounds of similar chemical or biologic composition to CSB-111.
2. Prior malignancy except for fully resected skin cancers.
3. Current treatment with systemic steroids, or immunosuppressive agents.
4. Known renal or hepatic disease.
5. Laboratory values:

   1. Leukocytes <3000/mcL
   2. Absolute neutrophil count <1500 mcL
   3. Platelets <100,000 mcL
   4. Total bilirubin >1.5 x Upper limit of normal (ULN)
   5. Aspartate Transaminase (AST)/ Alanine Aminotransferase (ALT) >2.5 x ULN
   6. Albumin <3.7 g/dL
   7. Gamma glutamyl transferase (GGT) >2.5 ULN
   8. eGFR <60 mL/min/1.73 m2 measured in the prior 30 days before administration of CSB-111
6. Having received any investigational product in the prior three months of receiving CSB-111.
7. Currently participating in any clinical trials, except observational studies.
8. Any acute or chronic inflammatory disease, autoimmune disorders, or medical conditions that in the investigator's opinion may interfere with the study procedures or the interpretation of the study results such as infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
9. Participants who have any condition that would prevent them from receiving a PET scan.
10. Female participants who are pregnant (confirmed via a positive serum or urine β-hCG test on the day of procedure prior to CSB-111 administration).
11. Female participants who are breastfeeding.
12. Unable or unwilling to use adequate contraception prior to study, during study participation and for one week post-injection for both females and males.
13. Any medical condition which, in the opinion of the investigator, may interfere with participation in the study and/or alter the biodistribution of CSB-111.
14. Mentally incapacitated or unable to understand the informed consent.
15. Participants who, in the opinion of the investigator, have underlying psychological conditions which may negatively impact their wellbeing if participating.
16. Prisoners.
17. Staff and family members of CytoSite.
18. Staff reporting to the principal investigator (PI).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Organ-level dosimetry of CSB-111 and total body and effective dose | PET/CT imaging up to 180 minutes post-injection
  milli-Sieverts [mSi]
Percentage of intact CSB-111 in blood samples up to 185 min after injection, using HPLC | From 65 to 185 minutes after injection
  Intact CSB-111 percentage in blood
Total radioactivity via gamma counter of cell pellet, plasma protein and unbound radioactivity in blood samples up to 65 min | Up to to 185 minutes post dose
  milli-Curies [mCi]
Concentration of intact CSB-111 in urine | up to 4 hours after injection or until below the level of detection
  Intact CSB-111 in urine in picograms
Percentage of intact CSB-111 in urine | up to 4 hours after injection or until below the level of detection
  Percentage of intact CSB-111 in urine compared to initial dose

SECONDARY OUTCOMES:
Overall AEs frequency and frequency per grade of AEs related to CSB-111 according to Medical Dictionary for Regulatory Activities (MedDRA)/ Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0 | up to 2 days post dose
  Overall AEs frequency and frequency per grade of AEs. All AE's in this study will be listed as an endpoint.

OTHER OUTCOMES:
Regional (organ) accumulation of CSB-111 | PET/CT imaging up to 180 minutes post-injection or until below limits of detection
  Dosimetry in organs in milli-Sieverts [mSi]

CONTACTS AND LOCATIONS:
Overall Officials: Colin Miller, Study Director — CytoSite Bio Inc.
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No